CLINICAL TRIAL: NCT04740775
Title: Clinical Study to Evaluate LiquiBand® Exceed™ and LiquiBand® Rapid™ for Closure of Surgical Incisions Associated With Abdominal Surgery
Brief Title: LiquiBand® Exceed™ and LiquiBand® Rapid™ for General Surgery Procedures
Acronym: Exceed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Collaborators: BioStat International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Exceed 01-2020
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Surgical Wound
Keywords: Topical Skin Adhesives,; Cyanoacrylate; LiquiBand Exceed; Wound Closure; LiquiBand Rapid
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: 2-arm, non-comparative, open-label, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LiquiBand Exceed (Experimental): Surgical wound closure using the LiquiBand Exceed Topical Skin Adhesive
  Interventions: Device: LiquiBand Exceed
- Liquiband Rapid (Experimental): Surgical wound closure using the LiquiBand Rapid Topical Skin Adhesive
  Interventions: Device: LiquiBand Rapid

INTERVENTIONS:
Device: LiquiBand Exceed — Cyanoacrylate glue for closure of surgical wounds
  Arms: LiquiBand Exceed
Device: LiquiBand Rapid — Cyanoacrylate glue for closure of surgical wounds
  Arms: Liquiband Rapid

SUMMARY:
The purpose of this post market study is to evaluate the performance and safety of LiquiBand® Exceed™ and LiquiBand® Rapid™ for closure of surgical incisions associated with abdominal surgery.

DETAILED DESCRIPTION:
LiquiBand® Exceed™ and LiquiBand® Rapid™ are the "study" devices. The study devices are an adhesive used to close surgical wounds. When the adhesive is applied to the skin, it polymerizes (forms a chemical bond) within minutes due to the moisture on the skin's surface and allows the wound edges to remain in the correct position. The use of the study devices are not "investigational" (experimental) because it is already cleared for doctors to use for surgical wound closure in the United States of America.

In this study, LiquiBand® Exceed™ and LiquiBand® Rapid™ will be used to close surgical wounds following general abdominal surgery. Subjects will be followed up for 14-days post surgery, and safety and performance of the study device will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of these criteria at time of enrollment may be included in the investigation:

1. Subject is ≥ 18 years of age
2. Subject is to undergo general abdominal surgery
3. Planned incision(s) are expected to be 4cm or greater in length
4. Subject is willing and able to comply with the protocol and follow up period
5. Subject is willing and able to give written informed consent

Exclusion Criteria:

Patients who meet any one of these criteria will be excluded from the study:

1. Subject is pregnant or nursing
2. Subject has inadequate or unsuitable tissue e.g. due to radiation damage, ulceration compromised vascularity, history of compromised wound heal.
3. Subject has a sensitivity to cyanoacrylates or formaldehyde
4. Subject has a known sensitivity to topical skin adhesives
5. Subject has active or potential infection at the surgical site
6. Subject has a history of keloid formation
7. Subject has a known vitamin C or zinc deficiency
8. Subject has a connective tissue disorder
9. Subject has uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of wound dehiscence | 14 days post-surgery
  Proportion of subjects with evidence of partial or complete dehiscence assessed by the investigator

SECONDARY OUTCOMES:
Safety of Liquiband Exceed, assessed by incidence of device-related AEs / SAEs | 14-days post-surgery
  Proportion of subjects who experience at least one device-related AE/SAE
Surgeon satisfaction with the device | Day 0
  To be assessed by the investigator using a Likert scale at the time of surgery
Cosmetic outcome | 14-days post-surgery
  Investigator assessment of wound cosmesis using the Modified Hollander Wound Evaluation Scale (HWES).
  This will be modified to a 6-point scale with one point assigned to any of the following observed wound appearances: step-off borders, contour irregularities, margin separation, edge inversion, excessive distortion, and overall appearance of wound. A HWES of 0 will indicate an optimal wound appearamce, with each point between 1 and 6 indicating a less adequate appearance of the wound.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Carbonnell, MD, Principal Investigator — Prisma Health-Upstate
Locations (3):
- United States (3):
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Prisma Health, Greenville, South Carolina
  - Prisma Health, Greer, South Carolina

IPD SHARING:
Plan to Share IPD: No